CLINICAL TRIAL: NCT07308405
Title: Comparative Clinical Evaluation of Coronally Advanced Flap With Platelet Rich Fibrin Membrane and Chorion Membrane in the Treatment of Human Gingival Recession
Brief Title: Evaluating Coronally Advanced Flap With Platelet-rich Fibrin Membrane and Chorion Membrane for Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dental Sciences, Bareilly, Uttar Pradesh, India (Other)
Responsible Party: Principal Investigator, Bimmi Tripathi, Doctor-primary Investigator, Institute of Dental Sciences, Bareilly, Uttar Pradesh, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDS/ETHCC/14/08
Record Dates: First submitted 2025-11-22; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Gingival Recession
Keywords: Coronally advanced flap; platelet rich fibrin; root coverage; chorion membrane; Gingival Recession Localized Moderate
MeSH Terms: conditions — Gingival Recession | interventions — Tissue Banks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental site A: patient were treated with coronally advanced flap and PRF (Experimental): Twenty five sites in each of 25 patient were treated with coronally advanced flap (CAF) and platelet-rich fibrin (PRF) membrane;
  Interventions: Procedure: Coronally advanced flap (CAF) with platelet-rich fibrin (PRF)
- Experimental site B: patient were treated with coronally advanced flap (CAF) and CM (Experimental): Twenty five sites in each of other 25 patient were treated with coronally advanced flap (CAF) and chorion membrane (CM)
  Interventions: Procedure: A similar surgical procedure was followed for the recipient bed preparation similar to that for the PRF membrane. A chorion membrane (Tissue bank, Tata Memorial Hospital, Mumbai, Maharashtra, India) o

INTERVENTIONS:
Procedure: Coronally advanced flap (CAF) with platelet-rich fibrin (PRF) — Description: After achieving adequate anaesthesia with 2% lignocaine (1:80,000 adrenaline), an intrasulcular incision was made on the buccal aspect of the involved teeth. Two horizontal incisions were placed from the mesial and distal angles to the papillae at the CEJ, without involving adjacent gingival margins. From their ends, two bevelled, slightly divergent oblique incisions were extended beyond the mucogingival junction, creating a trapezoidal flap. A full-thickness flap was raised up to the MGJ, followed by split-thickness dissection apically, with periosteal release to allow passive coronal mobilization. Adequate mobilization was defined as the flap margin reaching passively coronal to the CEJ. The coronal papilla soft tissue was de-epithelialized to prepare connective tissue beds for suturing of the coronally advanced flap. At the recipient site, the prepared PRF membrane was placed over the denuded root surfaces.
  Arms: Experimental site A: patient were treated with coronally advanced flap and PRF
Procedure: A similar surgical procedure was followed for the recipient bed preparation similar to that for the PRF membrane. A chorion membrane (Tissue bank, Tata Memorial Hospital, Mumbai, Maharashtra, India) o
  Arms: Experimental site B: patient were treated with coronally advanced flap (CAF) and CM

SUMMARY:
The present study was a double-blind, randomised, controlled clinical trial with a parallel design, comparing the coronally advanced flap (CAF) with platelet-rich fibrin (PRF) and chorion membrane (CM) for the treatment of isolated gingival recession defects. A total of 50 patients were randomly divided into; Experimental site A: Twenty five sites were treated with coronally advanced flap (CAF) and platelet-rich fibrin (PRF) membrane; Experimental site B: Twenty five sites were treated with coronally advanced flap (CAF) and chorion membrane (CM)The study was conducted in accordance with the Declaration of Helsinki, protocol was developed and ethical clearance was obtained from the Institutional Ethics Committee, Institute of Dental Sciences, Bareilly, India [IDS/ETHCC/14/08]. As per protocol, a study was conducted in five phases: (1) initial screening; (2) initial therapy and clinical measurements; (3) surgical therapy; (4) maintenance phase; and (5) post-operative evaluation after 1 month, 3 months, and 6 months.

DETAILED DESCRIPTION:
Platelet-rich fibrin (PRF), a second-generation platelet concentrate, accelerates soft and hard tissue regeneration. Chorion membrane, of fetal origin, has wound-modulating properties. This study aimed to evaluate and compare the clinical outcomes of PRF and chorion membrane in treating isolated Miller's Class I or II gingival recession defects. Fifty recession defects in 50 patients were randomly treated with a coronally advanced flap (CAF) and PRF membrane (site A, n = 25) or CAF with chorion membrane (site B, n = 25). Clinical parameters recorded at baseline, 1, 3, and 6 months included recession depth (RD), recession width (RW), clinical attachment level (CAL), width of keratinised gingiva (WKG), plaque index (PI), gingival index (GI), and gingival biotype. Statistical analysis compared outcomes across follow-up intervals. At six months, both groups demonstrated significant improvements in RD, RW, CAL, WKG, PI, and GI compared with baseline. Mean percentage root coverage was 86.76 ± 13.76 in the PRF group and 82.89 ± 15.65 in the chorion group, with no statistically significant difference between them. Sites with an initial thin biotype showed conversion to a thick biotype in both groups. Both PRF and chorion membrane demonstrated predictable effectiveness for managing isolated recession defects, with comparable outcomes. Longitudinal studies are needed to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-35 years
* In good general health
* Isolated Miller's Class I or II gingival recession ≥ 2 mm
* ≥ 1 mm keratinised tissue apical to root exposure
* Identifiable CEJ (cementoenamel junction)

Exclusion Criteria:

* Poor oral hygiene after Phase I therapy
* Smoking or alcohol use
* Occlusal disharmony
* Parafunctional habits
* Non-vital or endodontically treated teeth
* Caries, restorations, or crowns at the CEJ
* Frenum pull at the attached gingiva
* Previous surgery in the area

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recession depth (RD) | Baseline, prior to surgery and at 1 month, 3 months and 6 months follow-up visits
  Measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin
Recession width (RW) | Baseline, prior to surgery and at 1 month, 3 months and 6 months follow-up visits
  Measured between mesial and distal papillae across the buccal surface at the CEJ level
Clinical attachment level (CAL) | Baseline, prior to surgery and at 1 month, 3 months and 6 months follow-up visits:
  Measured from the CEJ to the bottom of the gingival sulcus;
Width of keratinized gingiva (WKG) | Baseline, prior to surgery and at 1 month, 3 months and 6 months follow-up visits
  Measured from the gingival margin to the mucogingival junction (MGJ)
Assessment of gingival biotype | Baseline, prior to surgery and at 1 month, 3 months and 6 months follow-up visits
  Evaluated based on the transparency of the probe through the gingival margin while probing the sulcus at the midfacial aspect of teeth

CONTACTS AND LOCATIONS:
Overall Officials: Shatyajit Naik, MDS, Study Chair — Institute of Dental Sciences, Bareilly, Uttar Pradesh, India
Locations (1):
- Department of Periodontics and implantology , Institute of Dental sciences, Bareilly, Uttar Pradesh, India, Bareilly, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
the clinical mesurement values were shared for statistical analysis
Supporting Information: SAP
Time Frame: it is completed
Access Criteria: statician will acess the information for statistical analysis

REFERENCES:
- [Background] Bertl K, Spineli LM, Mohandis K, Stavropoulos A. Root coverage stability: A systematic overview of controlled clinical trials with at least 5 years of follow-up. Clin Exp Dent Res. 2021 Oct;7(5):692-710. doi: 10.1002/cre2.395. Epub 2021 Feb 9. PMID 33565266
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Derived] Tripathi B, Manjunath RGS, Garg J, Gokhale ST, Nagate RR, Nishant K, Al-Qahtani SM, Al Magbol M, Tikare S, Chaturvedi M, Al-Qarni MA, Elagib MFA, Javali MA, Chaturvedi S. PRF membrane vs. chorion membrane with coronally advanced flap: a clinical study on gingival recession. Odontology. 2026 Jan 17. doi: 10.1007/s10266-026-01312-8. Online ahead of print. PMID 41545633

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT07308405/Prot_SAP_ICF_000.pdf